CLINICAL TRIAL: NCT01736618
Title: Subcutaneous Implantable Cardioverter Defibrillator (S-ICD®) System Post Approval Study
Brief Title: S-ICD® System Post Approval Study
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BSC CRM CDM00055718; BSC CRM CDM00055718 (Registry Identifier: S-ICD® PAS)
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-06

CONDITIONS: Primary Prevention of Sudden Cardiac Arrest; Secondary Prevention of Sudden Cardiac Arrest
Keywords: subcutaneous implantable defibrillator, post approval study, sudden cardiac arrest, Cameron Health defibrillator
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- S-ICD System Implant Attempt: All participants undergo an S-ICD System Implant attempt.
  Interventions: Device: S-ICD System

INTERVENTIONS:
Device: S-ICD System

SUMMARY:
The purpose of the S-ICD Post Approval Study is to document long term safety and effectiveness outcomes associated with the implantation of the SQ-RX pulse generator and Q-TRAK electrode in a commercial clinical setting.

DETAILED DESCRIPTION:
The S-ICD Post Approval Study is a non-randomized registry that will retrospectively enroll subjects who participated in the S-ICD Clinical Investigation (IDE G090013) and prospectively enroll new candidates for the S-ICD System. The target enrollment sample size is 1,616 subjects at up to 150 investigational sites to achieve 1,025 subjects in the analysis cohort at 60 months.

* The primary safety endpoint of the study is the Type I (caused by the S-ICD System) Complication Free Rate at 60 months compared to a performance goal of 85%.
* The primary effectiveness endpoint is the Overall Shock Effectiveness in Converting Spontaneous Discrete Episodes of ventricular tachycardia /ventricular fibrillation (VT/VF) through 60 months compared to a performance goal of 94%.
* The secondary safety endpoint of the study is the Electrode-Related Complication Free Rate at 60 months compared to a performance goal of 92.5%.
* The secondary effectiveness endpoint is First Shock Effectiveness in Converting Induced (Acute) and Spontaneous Discrete Episodes of VT/VF through 60 months compared to a performance goal of 84.0%.

Additional objectives include characterization of long term safety and effectiveness in subjects of varied body habitus and in traditionally underrepresented populations.

Subjects must meet the following criteria to be eligible for inclusion in the study:

1. Eligible for implantation with an S-ICD System, OR previously implanted with an S-ICD System in the S-ICD System Clinical Investigation (IDE G090013)
2. Willing and able to provide written informed consent or have informed consent provided by a legal representative

Subjects who meet the following criteria must be excluded from the study:

1. Remaining life expectancy of less than 360 days

Enrolled subjects will be followed at the implant procedure, pre-discharge and annual (±60 days) follow-up visits. Subjects are followed according to the standard of care at their participating investigational center.

The primary and secondary safety and effectiveness endpoints will include a compilation of S-ICD IDE study and S-ICD PAS study subject data

ELIGIBILITY:
Inclusion Criteria:

* Eligible for implantation with an S-ICD System, OR previously implanted with an S-ICD System in the S-ICD System Clinical Investigation (IDE G090013)

AND

* Willing and able to provide written informed consent or have informed consent provided by a legal representative

Exclusion Criteria:

* Remaining life expectancy of less than 360 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The S-ICD System is intended to provide defibrillation therapy for the treatment of life-threatening ventricular tachyarrhythmias in patients who do not have symptomatic bradycardia, incessant ventricular tachycardia, or spontaneous, frequently recurring ventricular tachycardia that is reliably terminated with anti-tachycardia pacing.
Sampling Method: Probability Sample
Enrollment: 1766 (Actual)
Dates: Start 2013-03-12 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Macuare-Gorden, MD, Study Director — Boston Scientific Corporation
Locations (87):
- United States (87):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Cardiovascular Associates of Mesa, Mesa, Arizona
  - Phoenix Cardiovascular Group, Phoenix, Arizona
  - Arizona Arrhythmia Consultants, PLC, Scottsdale, Arizona
  - PIMA Heart Physicians, PC, Tucson, Arizona
  - St. Vincent Heart Clinic Arkansas, Little Rock, Arkansas
  - Providence St. Joseph Medical Center, Burbank, California
  - Sequoia Hospital, East Palo Alto, California
  - Sharp Grossmont Hospital, El Cajon, California
  - California Heart Associates, Fountain Valley, California
  - University of California San Diago, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Huntington Memorial Hospital/Foothill Cardiology, Pasadena, California
  - Sharp Memorial Hospital, San Diego, California
  - St. John's Health Center, Santa Monica, California
  - Memorial Medical Center (UCH-MHS), Colorado Springs, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Cardiac Arrhythmia Services, Inc, Fort Lauderdale, Florida
  - St. Vincent's Ambulatory Care (Jacksonville, FL), Jacksonville, Florida
  - James A Haley Veterans Affairs Hospital, Tampa, Florida
  - University Community Hospital (Florida Hospital)/Advent Health Tampa, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University Hospital (Augusta, GA), Augusta, Georgia
  - Augusta University, Augusta, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - St. Joseph Hospital, Savannah, Georgia
  - CorVita Science Foundation, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Advocate Health and Hospitals Corporation/Midwest Heart Foundation, Lombard, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Indiana University -Ball, Muncie, Indiana
  - St. Luke's Unity Point, Cedar Rapids, Iowa
  - Norton Audobon Hospital, Louisville, Kentucky
  - Union Memorial Hospital, Baltimore, Maryland
  - John's Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hosptial, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mid-America Heart Institute - St. Luke's Hospital, Kansas City, Missouri
  - Cox Health Center for Research and Innovation, Springfield, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Bergen Cardiology, Omaha, Nebraska
  - Catholic Medical Center, Manchester, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Our Lady of Lourdes Medical Center, Haddon Heights, New Jersey
  - Jersery Shore Medical Center, Neptune City, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Albany Medical Center, Albany, New York
  - Maimonides Hospital, Brooklyn, New York
  - Beth Israel Medical Center, New York, New York
  - Mount Sinai, New York, New York
  - Stonybrook University Medical Center, Stony Brook, New York
  - Novant Health Heart and Vascular, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Summa Health, Akron, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - University Hospital Cleveland, Cleveland, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Ohio Health Research, Columbus, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Lake West Hospital, Willoughby, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Heart Center, Columbia, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - HeartPlace Mid-Cities EP, Bedford, Texas
  - North Texas Heart Center, Dallas, Texas
  - Univeristy of Texas Health Science Center, The Woodlands, Texas
  - University of Utah Hospital and Clinic, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Fairfax, Falls Church, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Hunter Holmes VA Medical Center, Richmond, Virginia
  - Virginia Cardiovascular Specialists, Richmond, Virginia
  - Virginia Commonwealth Univeristy, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Kootenai Heart Clinics, Spokane, Washington
  - The Vancouver Clinic, Vancouver, Washington
  - St. Mary's Hospital, Huntington, West Virginia

REFERENCES:
- [Derived] Weiss R, Knight BP, El-Chami M, Aasbo J, Hanon S, Sadhu A, Sidhu M, Brisben AJ, Carter N, Burke MC, Gold M. Impact of Age on Subcutaneous Implantable Cardioverter-Defibrillator in a Large Patient Cohort: Mid-Term Follow-Up. JACC Clin Electrophysiol. 2023 Oct;9(10):2132-2145. doi: 10.1016/j.jacep.2023.06.013. Epub 2023 Sep 6. PMID 37676200
- [Derived] Gold MR, El-Chami MF, Burke MC, Upadhyay GA, Niebauer MJ, Prutkin JM, Herre JM, Kutalek S, Dinerman JL, Knight BP, Leigh J, Lucas L, Carter N, Brisben AJ, Aasbo JD, Weiss R; S-ICD System Post Approval Study Investigators. Postapproval Study of a Subcutaneous Implantable Cardioverter-Defibrillator System. J Am Coll Cardiol. 2023 Aug 1;82(5):383-397. doi: 10.1016/j.jacc.2023.05.034. PMID 37495274
- [Derived] Gold MR, Aasbo JD, Weiss R, Burke MC, Gleva MJ, Knight BP, Miller MA, Schuger CD, Carter N, Leigh J, Brisben AJ, El-Chami MF. Infection in patients with subcutaneous implantable cardioverter-defibrillator: Results of the S-ICD Post Approval Study. Heart Rhythm. 2022 Dec;19(12):1993-2001. doi: 10.1016/j.hrthm.2022.07.031. Epub 2022 Aug 6. PMID 35944889
- [Derived] Burke MC, Aasbo JD, El-Chami MF, Weiss R, Dinerman J, Hanon S, Kalahasty G, Bass E, Gold MR. 1-Year Prospective Evaluation of Clinical Outcomes and Shocks: The Subcutaneous ICD Post Approval Study. JACC Clin Electrophysiol. 2020 Nov;6(12):1537-1550. doi: 10.1016/j.jacep.2020.05.036. Epub 2020 Aug 26. PMID 33213814
- [Derived] El-Chami MF, Burke MC, Herre JM, Shah MH, Sadhu A, Niebauer MJ, Kutalek SP, Carter N, Gold MR. Outcomes of subcutaneous implantable cardioverter-defibrillator in dialysis patients: Results from the S-ICD post-approval study. Heart Rhythm. 2020 Sep;17(9):1566-1574. doi: 10.1016/j.hrthm.2020.04.036. Epub 2020 May 4. PMID 32376304
- [Derived] Gold MR, Aasbo JD, El-Chami MF, Niebauer M, Herre J, Prutkin JM, Knight BP, Kutalek S, Hsu K, Weiss R, Bass E, Husby M, Stivland TM, Burke MC. Subcutaneous implantable cardioverter-defibrillator Post-Approval Study: Clinical characteristics and perioperative results. Heart Rhythm. 2017 Oct;14(10):1456-1463. doi: 10.1016/j.hrthm.2017.05.016. Epub 2017 May 11. PMID 28502872

RESULTS

PARTICIPANT FLOW:
Groups:
- S-ICD System Implant Attempt: All subjects undergo an S-ICD System implant procedure.
Period: Overall Study
Arm/Group | S-ICD System Implant Attempt
Started | 1766
Completed | 767
Not Completed | 999
Not completed — Death | 294
Not completed — Lost to Follow-up | 193
Not completed — Withdrawal by Subject | 54
Not completed — Subject unable to be followed at study location | 223
Not completed — Physician Decision | 33
Not completed — Transplant or removal of target organ | 19
Not completed — Change in indication or condition | 78
Not completed — Study device explant | 103
Not completed — Unable to complete implant | 2

BASELINE CHARACTERISTICS:
Population: All subjects who received an implant attempt are included.
Arm/Group | S-ICD System Implant Attempt
Number analyzed (Participants) | 1766
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 542
  Male | 1224
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: Caucasian | 1048
  Race and Ethnicity: Black, of African heritage | 508
  Race and Ethnicity: Hispanic or Latino | 104
  Race and Ethnicity: Asian | 22
  Race and Ethnicity: American Indian or Alaska Native | 16
  Race and Ethnicity: Native Hawaiian or other Pacific Islander | 8
  Race and Ethnicity: Other | 5
  Race and Ethnicity: Multi-racial | 9
  Race and Ethnicity: Not Disclosed | 46
Region of Enrollment [Number; unit: participants]
  United States | 1766
Device Indication [Count of Participants; unit: Participants]
  Primary prevention | 1359
  Secondary prevention | 407
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: % of LV volume ejected per heart beat] — Population: EF was only available for 1714 participants.
  % of LV volume ejected per heart beat
    number analyzed (Participants) | 1714
    (all) | 32.3 (14.6)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI was only available for 1762 participants
  kg/m^2
    number analyzed (Participants) | 1762
    (all) | 29.9 (7.6)
History of Atrial Fibrillation [Count of Participants; unit: Participants] — Population: Atrial Fibrillation was only available for 1760 participants.
  Participants
    number analyzed (Participants) | 1760
    (all) | 732
History of Hypertension [Count of Participants; unit: Participants] — Population: Hypertension was only available for 1760 participants.
  Participants
    number analyzed (Participants) | 1760
    (all) | 1089
History of Diabetes [Count of Participants; unit: Participants] — Population: Diabetes history was only available for 1760 participants.
  Participants
    number analyzed (Participants) | 1760
    (all) | 592
History of Myocardial Infarction [Count of Participants; unit: Participants] — Population: History of Myocardial Infarction was only available for 1737 participants.
  Participants
    number analyzed (Participants) | 1737
    (all) | 582
History of Kidney Disease [Count of Participants; unit: Participants] — Population: History of Kidney Disease was only available for 1760 participants.
  Participants
    number analyzed (Participants) | 1760
    (all) | 432
Creatinine Level [Mean (Standard Deviation); unit: mg/dL] — Population: Creatinine level was only available for 1629 participants.
  mg/dL
    number analyzed (Participants) | 1629
    (all) | 1.8 (2.2)
History of Cancer [Count of Participants; unit: Participants] — Population: History of Cancer was only available for 1760 participants.
  Participants
    number analyzed (Participants) | 1760
    (all) | 28
History of Coronary Artery Bypass Graft (CABG) [Count of Participants; unit: Participants] — Population: History of CABG was only available for 1752 participants.
  Participants
    number analyzed (Participants) | 1752
    (all) | 284
History of Percutaneous Revascularization [Count of Participants; unit: Participants] — Population: History of Percutaneous Revascularization was only available for 1744 participants.
  Participants
    number analyzed (Participants) | 1744
    (all) | 484

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Free From Type I Complication
Description: Type I complications are adverse events caused by a component of the S-ICD System (i.e. pulse generator, electrode, EIT or programmer) that results in permanent loss of device function, invasive intervention or death.
Time Frame: 60 months (1800 days)
Population: S-ICD PAS enrolled de novo implant subjects as well as prior IDE participants. Primary Safety endpoint includes subjects enrolled in S-ICD PAS combined with the subjects from the S-ICD IDE (NCT# 01064076). S-ICD PAS had 1643 de novo implant attempts and 123 prior IDE implant subjects, for endpoint analyses this was combined with the data from the 198 IDE implant attempt subjects that did not participate in S-ICD PAS, totaling 1964 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | S-ICD System Implant Attempt
Number analyzed (Participants) | 1964
Participants | 1869
Statistical Analysis 1: Comparison: S-ICD System Implant Attempt; Ho: The Type I Complication Free Rate at 60 months (p1) does not exceed the performance goal of 85.0%. Ho: p1 ≤ 85.0% Ha: The Type I Complication Free Rate at 60 months (p1) does exceed the performance goal of 85.0%. Ha: p1 > 85.0% The null hypothesis will be rejected if the lower one-sided 95% confidence bound of the proportional means model estimate, using the Peto method for standard error, exceeds the performance goal of 85.0%; Test type: Other; Kaplan-Meier = 92.9, 95% CI 1-sided [lower limit 91.4]

2. Primary Outcome: Overall Shock Effectiveness in Converting Spontaneous Discrete Episodes of VT/VF
Description: Overall shock effectiveness refers to conversion of an episode following on any of the 5 shocks (maximum) that may be delivered during a single episode. Discrete episodes of VT/VF are those that are temporally independent (<3 within a 24 hour period), unlike storm episodes, which occur in clusters (≥3 episodes within a 24 hour period). Episodes that spontaneously terminate will be excluded from this endpoint since the effectiveness of the shock cannot be evaluated in such circumstances.
Time Frame: 60 months (1825 days)
Population: Primary effectiveness endpoint includes subjects in S-ICD PAS combined with the subjects from the S-ICD IDE (NCT# 01064076). S-ICD PAS had 1637 de novo implants and 123 prior IDE implant subjects, for endpoint analyses this was combined with the data from the 191 IDE implanted subjects that did not participate in S-ICD PAS, totaling 1951 subjects. This endpoint analyzes all appropriate shocks.
Measure: Number; unit: S-ICD Shocks
Units Other Than Participants: S-ICD Shocks
Arm/Group | S-ICD System Implant Attempt
Number analyzed (Participants) | 1951
Number analyzed (S-ICD Shocks) | 512
S-ICD Shocks | 505
Statistical Analysis 1: Comparison: S-ICD System Implant Attempt; Ho: Overall Shock Effectiveness in Converting Spontaneous Discrete Episodes of VT/VF through 60 months (p1) does not exceed the performance goal of 94.0%. Ho: p1 ≤ 94.0% Ha: Overall Shock Effectiveness in Converting Spontaneous Discrete Episodes of VT/VF through 60 months (p1) does exceed the performance goal of 94.0%. Ha: p1 >94.0% The null hypothesis will be rejected if the lower one-sided 95% exact confidence bound of the estimate exceeds the performance goal of 94.0%; Test type: Other; Clopper-Pearson exact confidence bound = 98.6, 95% CI 1-sided [lower limit 97.4]

3. Secondary Outcome: Number of Participants Free From Electrode-related Complications
Description: The electrode related complications analyzed for this end-point include: complications occurring less than or equal to 30 days post implant that are attributable to structural electrode failure for electrode movement, electrode impendence out of range, electrode conductor fracture, deformation or breakage or insulation failure; OR occurring greater than 30 days post implant regardless of structural failure for electrode movement, electrode impendence out of range, electrode conductor fracture, deformation/breakage or insulation failure; OR occurring greater than 30 days post implant attributable to structural electrode failure for incomplete/improper header connection, in-subject damage to electrode, electrode revision to optimize therapy, electrode movement, infection, oversensing/undersensing. Additionally, a complication is an adverse event that results in permanent loss of device function, invasive intervention or death.
Time Frame: 60 months (1800 days)
Population: Secondary safety endpoint includes subjects in S-ICD PAS combined with the subjects from the S-ICD IDE (NCT# 01064076). S-ICD PAS had 1643 de novo implant attempts and 123 prior IDE implant subjects, for endpoint analyses this was combined with the data from the 198 IDE implant attempt subjects that did not participate in S-ICD PAS, totaling 1964 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | S-ICD System Implant Attempt
Number analyzed (Participants) | 1964
Participants | 1953
Statistical Analysis 1: Comparison: S-ICD System Implant Attempt; Ho: The Electrode-Related Complication Free Rate at 60 months (p1) does not exceed the performance goal of 92.5%. Ho: p1 ≤ 92.5% Ha: The Electrode-Related Complication Free Rate at 60 months (p1) does exceed the performance goal of 92.5%. Ha: p1 > 92.5% The null hypothesis will be rejected if the lower one-sided 95% confidence bound of the proportional means model estimate, using the Peto method for standard error, exceeds the performance goal of 92.5%; Test type: Other; Kaplan-Meier = 99.2, 95% CI 1-sided [lower limit 98.8]

4. Secondary Outcome: First Shock Effectiveness in Converting Induced (Acute) and Spontaneous Discrete Episodes of VT/VF
Description: The rate in first shock effectiveness in converting induced (acute) and spontaneous discrete episodes of VT/VF through 60 months (1825 days) is calculated as the number of successful first shock conversions divided by the total evaluable episodes Acute Tests included: S-ICD PAS Study: Acute tests include induced episodes during the initial implant hospitalization after enrollment. Inductions may have been done on different days, but all occurred before the patient was discharged after initial implant; IDE Study : Acute tests included induced episodes occurring during the initial implant procedure as well as subsequent hospitalization until the final system position was obtained.
  * Acute Test Shock Energy Levels included all energy levels in the PAS Study and only 65 Joule shocks in the IDE Study.
  * Acute Test Arrhythmias included all VT and VF episodes for the PAS Study and only VF episodes for the IDE Study.
Time Frame: 60 months (1825 days)
Population: The secondary effectiveness endpoint includes subjects in S-ICD PAS combined with the subjects from the S-ICD IDE (NCT# 01064076). S-ICD PAS had 1637 de novo implants and 123 prior IDE implant subjects, for endpoint analyses this was combined with the data from the 191 IDE implanted subjects that did not participate in S-ICD PAS, totaling 1951 subjects. This endpoint analyzes all induced (acute) or spontaneous appropriately treated discrete VT/VF shocks.
Measure: Number; unit: S-ICD Shocks
Units Other Than Participants: S-ICD Shocks
Arm/Group | S-ICD System Implant Attempt
Number analyzed (Participants) | 1951
Number analyzed (S-ICD Shocks) | 2195
S-ICD Shocks | 2071
Statistical Analysis 1: Comparison: S-ICD System Implant Attempt; Ho: The 1st Shock Effectiveness in Converting Induced (Acute) & Spontaneous Discrete VT/VF Episodes to 60 months (p1) does not exceed the performance goal of 84.0%. Ho: p1 ≤ 84.0% Ha: The 1st Shock Effectiveness in Converting Induced (Acute) & Spontaneous Discrete VT/VF Episodes to 60 months (p1) does exceed the performance goal of 84.0%. Ha: p1 >84.0% The null hypothesis will be rejected if lower one-sided 95% exact confidence bound of the estimate exceeds the performance goal of 84.0%; Test type: Other; Clopper-Pearson exact confidence bound = 94.4, 95% CI 1-sided [lower limit 93.5]

ADVERSE EVENTS:
Time Frame: Data was collected over a 60 month (5-year) follow-up period
Arm/Group | S-ICD System Implant Attempt
All-Cause Mortality (participants affected / at risk) | 294/1766
Serious Adverse Events (participants affected / at risk) | 638/1766
Other Adverse Events (participants affected / at risk) | 247/1766
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-ICD System Implant Attempt (N=1766)
Heart Failure (HF)/ Worsening HF (Cardiac disorders) | 63 (68)
Worsening VT/VF (Cardiac disorders) | 50 (55) — Worsening Ventricular Tachycardia/Ventricular Fibrillation - Cardiovascular related
Chest Pain - Cardiovascular related (Cardiac disorders) | 25 (26)
Cardiac Arrest (Cardiac disorders) | 25 (25)
Atrial Fibrillation / Atrial Flutter (Cardiac disorders) | 23 (24)
Bradycardia/ AV Block (Cardiac disorders) | 21 (21)
Pulseless Electrical Activity (PEA) (Cardiac disorders) | 20 (20)
Cardiogenic Shock (Cardiac disorders) | 15 (16)
Other -Cardiovascular related (Cardiac disorders) | 8 (8)
Palpitations (Cardiac disorders) | 2 (2)
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 2 (2)
Supraventricular Tachycardia (SVT) (Cardiac disorders) | 2 (2)
Angina (Cardiac disorders) | 1 (1)
Aortic Stenosis (Cardiac disorders) | 1 (1)
Inflammation - Cardiovascular related (Cardiac disorders) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 6 (8)
Multisystem Failure - Other (General disorders) | 53 (53)
Death - unknown cause (General disorders) | 38 (38)
Syncope - Cardiovascular (Cardiac disorders) | 11 (12)
Near Syncope/Dizziness/Shortness of Breath/Confusion (Cardiac disorders) | 2 (2)
Syncope - Non-cardiovascular (General disorders) | 7 (8)
Chest pain - Non-cardiac other (General disorders) | 6 (7)
Abnormal Laboratory Values (General disorders) | 4 (5)
Multiple Symptoms (General disorders) | 2 (2)
Near Syncope/Dizziness/Shortness of Breath/Confusion (General disorders) | 1 (1) — Non-Cardiovascular
Other - Patient Condition - Non-cardiovascular (General disorders) | 1 (1)
Infection - Non-device/procedure related (Infections and infestations) | 49 (51)
Infection - S-ICD System/Implant Procedure related (Injury, poisoning and procedural complications) | 45 (45)
Hematoma <= 30 days post-implant - Procedure related (Injury, poisoning and procedural complications) | 12 (12)
Infection - Incisional/Superficial Infection - Procedure related (Injury, poisoning and procedural complications) | 10 (10)
Adverse Reaction - Hypotension - Procedure related (Injury, poisoning and procedural complications) | 9 (9)
Discomfort - Post-op > 30-Days - Device related (Product Issues) | 5 (5)
Sub-optimal Electrode Position - Procedure related (Injury, poisoning and procedural complications) | 4 (4)
Adverse Reaction to Medications - Procedure related (Injury, poisoning and procedural complications) | 3 (3)
Elective Device Replacement (Injury, poisoning and procedural complications) | 3 (3) — Replacement of the S-ICD
Electrode Movement - Procedure related (Injury, poisoning and procedural complications) | 3 (3)
Inadequate healing of incision site - Procedure related (Injury, poisoning and procedural complications) | 3 (3)
Trauma - Other (Injury, poisoning and procedural complications) | 3 (3) — Non-device system related trauma
Cardiac arrest - Procedure related (Injury, poisoning and procedural complications) | 2 (2)
Electrode movement - Electrode related (Product Issues) | 2 (2)
Respiratory Failure - Procedure related (Injury, poisoning and procedural complications) | 2 (2)
Adverse Reaction Respiratory - Procedure Related (Injury, poisoning and procedural complications) | 1 (1)
Bleeding - Procedure related (Injury, poisoning and procedural complications) | 1 (1)
Fever - Procedure related (Injury, poisoning and procedural complications) | 1 (1)
Heart Failure / Worsening of Heart Failure - Procedure related (Injury, poisoning and procedural complications) | 1 (1)
Hematoma - Pocket (> 30 days post-implant) (Injury, poisoning and procedural complications) | 1 (1)
Hematoma > 30 days post-implant - Procedure related (Injury, poisoning and procedural complications) | 1 (1)
PG movement / Revision - Other (Injury, poisoning and procedural complications) | 1 (1)
Pleural Effusion - Procedure related (Injury, poisoning and procedural complications) | 1 (1)
Pneumothorax - Procedure related (Injury, poisoning and procedural complications) | 1 (1)
Pulseless Electrical Activity (PEA) Post Anesthesia prior to Implant (Injury, poisoning and procedural complications) | 1 (1)
Seroma - Procedure related (Injury, poisoning and procedural complications) | 1 (1)
Sub-optimal device and electrode position - Procedure related (Injury, poisoning and procedural complications) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (15)
Neurological (Nervous system disorders) | 1 (1)
Inappropriate Shock - Inappropriate Sensing: Cardiac Oversensing (Product Issues) | 57 (64)
Inappropriate Shock - Inappropriate Sensing: Extra-cardiac Oversensing (Product Issues) | 12 (13)
Inappropriate Shock - Above Programmed Rate Zone (Product Issues) | 11 (12)
Premature Cell Battery Depletion (Product Issues) | 11 (11)
Inappropriate Shock - Inappropriate Sensing: Discrimination Error (Product Issues) | 6 (8)
Unable to Convert - During Device System Implant Procedure (Product Issues) | 6 (7)
Erosion - Device related (Product Issues) | 6 (6)
Appropriate Shock - Accelerated Arrhythmia (Product Issues) | 1 (1)
Electrode Conductor Fracture- Presumed Twiddler's Syndrome (Product Issues) | 1 (1)
Erosion - Electrode related (Product Issues) | 1 (1)
Erosion - Imminent Erosion - Device related (Product Issues) | 1 (1)
Inability to Communicate with the Device (Product Issues) | 1 (1)
Inappropriate Shock - Inappropriate Sensing: Baseline Shift (Product Issues) | 1 (1)
Trauma to Device (Product Issues) | 1 (1)
Unable to Convert - During Device Testing Procedure >150 days - Patient condition (Product Issues) | 1 (1)
Undersensing - Device related (Product Issues) | 1 (1)
Psychological Disorder (Psychiatric disorders) | 4 (4)
Kidney Disease (Renal and urinary disorders) | 12 (12)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Shortness of Breath/Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myocardial Infarction (Vascular disorders) | 29 (30)
Stroke (Vascular disorders) | 24 (24)
Coronary Artery Disease (Vascular disorders) | 9 (9)
Bleeding - Other (Vascular disorders) | 4 (4)
Stroke - Procedure related (Injury, poisoning and procedural complications) | 4 (4)
Thrombosis (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 2 (3)
Peripheral Vascular Disease (Vascular disorders) | 2 (3)
Pulmonary Embolism (Vascular disorders) | 3 (3)
Transient Ischemic Attack (TIA) (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 1 (1)
Discomfort - Post-op ≤ 30-Days - Procedure related (Injury, poisoning and procedural complications) | 10 (10)
Discomfort - Post-op ≤ 30-Days - Device related (Product Issues) | 2 (2)
Device Movement - Revision (Product Issues) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-ICD System Implant Attempt (N=1766)
Inappropriate Shock - Inappropriate Sensing: Cardiac Oversensing (Product Issues) | 109 (134)
Inappropriate Shock - Inappropriate Sensing: Extra-cardiac Oversensing (Product Issues) | 46 (47)
Discomfort - Post-op > 30-Days - Device related (Product Issues) | 25 (25)
Incisional/Superficial Infection - Procedure related (Injury, poisoning and procedural complications) | 24 (24)
Hematoma <= 30 days post-implant - Procedure related (Injury, poisoning and procedural complications) | 21 (21)
Discomfort - Post-op ≤ 30-Days - Procedure related (Injury, poisoning and procedural complications) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit publication to Sponsor for review at least 60 days prior to submission. Sponsor reserves the right to delete any confidential info or other proprietary info of Sponsor (not incl. Results). Sponsor may extend 90 days to protect its intellectual property (IP) interests. PI shall be free to publish the results of the study after: Initial Publication is published; notification by Sponsor that Initial Publication is no longer planned; or 12 mo. after the expiration date at all sites

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT01736618/Prot_SAP_000.pdf